CLINICAL TRIAL: NCT06536283
Title: Opiophobia in Postsurgical Adults With Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Sigma Theta Tau International (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0315; NCI-2024-06535 (Other: NCI-CTRP)
Record Dates: First submitted 2024-07-31; First posted 2024-08-02 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Opiophobia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Opiophobia in Postsurgical Adults: Participants that agree to take part in this study, partiicpants will have a virtual visit, via Zoom, about 7 days after you are discharged from the hospital. The visit will take about 20 minutes, and you will meet with a member of the research team to complete several questionnaires.
  Interventions: Other: 13-item Barriers Questionnaire (BQ-13); Other: Four-item Medication Adherence Questionnaire; Other: 14-item Hospital Anxiety and Depression Scale (HADS)

INTERVENTIONS:
Other: 13-item Barriers Questionnaire (BQ-13) — Given by questionnaire
Other: Four-item Medication Adherence Questionnaire — Given by questionnaire
Other: 14-item Hospital Anxiety and Depression Scale (HADS) — Given by questionnaire

SUMMARY:
To learn how people who underwent surgery feel about their prescribed opioid medication after they leave the hospital.

DETAILED DESCRIPTION:
To explore the barriers and fears related to use of opioids among a population of adults who underwent surgery for cancer who were prescribed opioids for home use during the first week following hospital discharge for a surgical treatment of a malignancy.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient with cancer admitted for cancer-related surgery
2. inpatient surgical hospital stay lasting at least 23 hours
3. discharged home with a prescription for opioid analgesics
4. able to read, speak, and consent in English.

Exclusion Criteria:

1. Age less than 18 years
2. not discharged with a prescription for opioid analgesia to manage pain
3. individuals for whom there is documentation of inability to provide consent in the medical record.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To explore the barriers and fears related to use of opioids among a population of adults who underwent surgery for cancer. | Through study completion, an average of 1 year.
  Use of opioids among a population of adults who underwent surgery for cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Eileen Hacker, PHD,RN, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The Univerisity of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org